CLINICAL TRIAL: NCT01904968
Title: Impact of Methylation Alterations in Colon Cancer: Epidemiology and Prognosis
Status: Withdrawn | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Piard PHRC K 2011
Record Dates: First submitted 2013-06-26; First posted 2013-07-22 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2013-07

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Colon cancers in patients living the Cote D'or area

SUMMARY:
We conducted a preliminary study in 2010 using the innovative Illumina GoldenGate (methylation assay) which has enabled us to characterize the level of methylation of 807 potential markers on a series of 200 adenocarcinomas of the colon (C18) and rectosigmoid junction (C19) resected between 1998 and 2001. The results, validated by pyrosequencing, allowed us to establish a panel of 12 markers to assess the level of methylation. The aim of this project is to validate the prognostic value of this panel in a second cohort of patients with adenocarcinomas (stage I to IV) resected between 2002 and 2006 in public and private hospitals (n=685).

This study relies on an original collection of surgical specimens of colorectal cancers resected in public and private hospitals among patients resident in the département of Côte-d'Or and followed by the cancer registry of Burgundy. Samples obtained from each cancer and from adjacent normal mucosa are stored in liquid nitrogen in the Ferdinand Cabane Biological Resources Centre(certified S 96900). Annotations are collected by the cancer registry staff from multiple sources (pathologists, gastroenterologists, oncologists and radiotherapists).

Pyrosequencing will be used to quantify the level of methylation. The percentage of methylated allele for each marker on cancerous DNA and the ratio of methylated markers to the number of markers analyzed will be determined. The molecular status of MSI, BRAF, KRAS, and PI3K will be taken into consideration.

To study the prognosis, relative and relapse free-survival will be calculated. A multivariate relative survival analysis will be performed to determine independent prognostic factors taking into account the characteristics of patients and tumours and epigenetic and molecular alterations. Epigenetic alterations will be described according to age group, sex and subsite. The epigenetic phenotypes will be evaluated according to already known molecular status using logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinomas of the colon (C18) and rectosigmoid junction (C19)
* Resident in Côte-d'Or
* Treated by surgical resection

Exclusion Criteria:

* Rectal cancer
* Cancer on Crohn's disease and ulcerate colitis
* Hereditary colon cancer (HNPCC, familial polyposis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colon cancers in patients living the Cote D'or area
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Quality control DNA | at baseline
Assessment of methylation level | at the baseline
MSI Phenotype evaluation | at the baseline
Mutational status evaluation of BRAF, KRAS and PI3KCA : | at the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Françoise PIARD, Principal Investigator — CHU Dijon /INSERM U866
Locations (1):
- CHU de Dijon, Dijon, France